CLINICAL TRIAL: NCT02994589
Title: A Comparison of OASIS Wound Matrix With Approved Dressings for Split Thickness Skin Graft Donor Sites
Brief Title: A Comparison of OASIS Wound Matrix With Approved Dressings for Skin Graft Donor Sites
Acronym: OASIS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was never started
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 5150267
Record Dates: First submitted 2015-08-31; First posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Skin Graft Complications
MeSH Terms: interventions — 2,4,6-tribromophenol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- OASIS® wound matrix (Experimental): OASIS wound matrix is a biologic extracellular matrix derived from porcine small intestine submucosa. Some components of OASIS wound matrix are similar to human dermis including types of collagens, elastin, glycoproteins and proteoglycans. In addition, OASIS wound matrix retains some growth factors that have been suggested to aid in the wound healing process. It is a FDA approved wound dressing indicated for use in a variety of ulcers, abrasions and surgical wounds.
  Interventions: Device: OASIS® wound matrix
- Tegaderm™(Absorbant, 3M) (Active Comparator): Transparent dressing allows for wound monitoring without changing the dressing Clear design takes the guesswork out of application over the wound Novel acrylic polymer pad technology designed to handle low to moderate wound drainage. No dressing breakdown in the wound. Low friction surface minimizes potential for friction and shear. Allows for gentle removal from skin. Barrier to external contaminants, body fluids, bacteria and viruses.
  Interventions: Other: Tegaderm™(Absorbant, 3M)
- Xeroform™ (Active Comparator): Xeroform™ Occlusive Petrolatum Gauze. 3% Bismuth Tribromophenate in a special petrolatum blend on fine mesh gauze. Non-adherent. Clings and conforms to all body contours.
  Interventions: Other: Xeroform™

INTERVENTIONS:
Other: Tegaderm™(Absorbant, 3M) — 3M™ Tegaderm™ Dressing helps provide the natural moisture balance conducive to wound healing.
  Arms: Tegaderm™(Absorbant, 3M)
Device: OASIS® wound matrix — OASIS® Matrix is indicated for the management of wounds including: partial- and full-thickness wounds, pressure ulcers, venous ulcers, chronic vascular ulcers, diabetic ulcers, trauma wounds (abrasions, lacerations, second-degree burns, skin tears), draining wounds, surgical wounds (donor sites/grafts, post-Mohs' surgery, post-laser surgery, podiatric, wound dehiscence).
  Arms: OASIS® wound matrix
Other: Xeroform™ — Xeroform™ consists of a fine-mesh gauze impregnated with bismuth tribromophenate.
  Arms: Xeroform™

SUMMARY:
The investigators objective is to compare OASIS wound matrix with other commonly used dressings available for the donor site in split thickness skin grafting in order to determine which dressing provides the best outcome based on pain level, time to healing and aesthetic outcome.

DETAILED DESCRIPTION:
Investigators seek to compare Oasis wound matrix with Tegaderm and Xeroform in order to determine whether advantages exist in one or more of the dressing types that are approved and currently used for split-thickness skin graft donor site dressings.

Patients will be randomly assigned to one of the three treatment groups and followed up post-operatively and treated as per current standard of care.

Data to be collected and analyzed includes: patient age, co-morbid illnesses, medication, skin-graft donor location, skin-graft donor area, STSG thickness, infection rate, complications involving the donor site, post-operative pain score every morning until hospital discharge, healing rate, photographs of the donor site immediately post-operatively and then at routine follow-up appointments.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo split thickness skin grafting
* patients able to consent without a proxy

Exclusion Criteria:

* confounding medical conditions
* previous skin grafting from site
* prior use of biological skin substitute on site

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Time to Heal | 7-21 days
  Patient will be followed up during routine post-operative appointments at the clinic weekly to check the healing process of the donor site wound.

SECONDARY OUTCOMES:
Aesthetic Outcome | 1-12 weeks
  During routine followup visits to the clinic, the donor site aesthetic outcome will be observed and recorded clinically and digitally (photographs). The Vancouver Scar Scale will be used.
Pain intensity measure | 7 days
  Self reported pain intensity in the morning and evening with activity over the past 7 days. Each item is scored on a scale of 0-10 (0= no pain, 10= highest intensity of pain)

CONTACTS AND LOCATIONS:
Overall Officials: Subhas Gupta, MD, PhD, Study Chair — Loma Linda University; Hahns Kim, MD, Principal Investigator — Loma Linda University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mostow EN, Haraway GD, Dalsing M, Hodde JP, King D; OASIS Venus Ulcer Study Group. Effectiveness of an extracellular matrix graft (OASIS Wound Matrix) in the treatment of chronic leg ulcers: a randomized clinical trial. J Vasc Surg. 2005 May;41(5):837-43. doi: 10.1016/j.jvs.2005.01.042. PMID 15886669
- [Result] Hankin CS, Knispel J, Lopes M, Bronstone A, Maus E. Clinical and cost efficacy of advanced wound care matrices for venous ulcers. J Manag Care Pharm. 2012 Jun;18(5):375-84. doi: 10.18553/jmcp.2012.18.5.375. PMID 22663170
- [Result] Eskes AM, Brolmann FE, Gerbens LA, Ubbink DT, Vermeulen H; REMBRANDT study group. Which dressing do donor site wounds need?: study protocol for a randomized controlled trial. Trials. 2011 Oct 17;12:229. doi: 10.1186/1745-6215-12-229. PMID 21999705
- [Result] Fernandes de Carvalho V, Paggiaro AO, Isaac C, Gringlas J, Ferreira MC. Clinical trial comparing 3 different wound dressings for the management of partial-thickness skin graft donor sites. J Wound Ostomy Continence Nurs. 2011 Nov-Dec;38(6):643-7. doi: 10.1097/WON.0b013e3182349d2f. PMID 22011820